CLINICAL TRIAL: NCT05127551
Title: A Prospective, Randomized, Controlled, Comparitive Multicenter Clinical Study of Glaukos® Trabecular Micro-Bypass System Model iS3 Infinite® vs Competitor in Adult Subjects With Primary Open-Angle Glaucoma (POAG)
Brief Title: Clinical Study of Glaukos® Trabecular Micro-Bypass System Model iS3 Infinite Vs. Competitor
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INFI-103-COMP
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma; Glaucoma, Open-Angle
Keywords: Glaucoma; MIGS
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iStent Infinite (Active Comparator): Subjects implanted with iStent Infinite system
  Interventions: Device: iStent Infinite
- Competitor Device (Active Comparator): Subject implanted with competitor device
  Interventions: Device: Competitor Device

INTERVENTIONS:
Device: iStent Infinite — Implantation of the iStent Infinite
  Arms: iStent Infinite
Device: Competitor Device — Implantation of competitor device
  Arms: Competitor Device

SUMMARY:
A study of the iStent Infinite product in the treatment of open-angle glaucoma vs competitor

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Open-Angle Glaucoma (POAG) or Secondary Pseudoexfoliative Glacoma (PEXG) or Secondary Pigmentary Glaucoma (PG)

Exclusion Criteria:

* Any other type of glaucoma including, but not limited to: traumatic glaucoma, angle recession glaucoma, uveitic glaucoma, neovascular glaucoma, angle closure glaucoma (ACG) and glaucoma associated with vascular disorders

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Diurnal Intraocular Pressure | Month 24
  Change in Mean Diurnal Intraocular Pressure from Baseline over time

CONTACTS AND LOCATIONS:
Locations (1):
- Glaukos Investigator Sites, Montreal, Qubec, Canada

REFERENCES:
- [Derived] Ahmed IIK, Berdahl JP, Yadgarov A, Reiss GR, Sarkisian SR Jr, Gagne S, Robles M, Voskanyan LA, Sadruddin O, Parizadeh D, Giamporcaro JE, Kothe AC, Katz LJ, Navratil T. Six-Month Outcomes from a Prospective, Randomized Study of iStent infinite Versus Hydrus in Open-Angle Glaucoma: The INTEGRITY Study. Ophthalmol Ther. 2025 May;14(5):1005-1024. doi: 10.1007/s40123-025-01126-x. Epub 2025 Mar 25. PMID 40128494